CLINICAL TRIAL: NCT06198335
Title: Comparison Of Modified Thoracoabdominal Nerve Block Through Perichondrial Approach and Transversus Abdominal Plane Block in Analgesia Efficacy And Recovery Quality Following Laparoscopic Cholecystectomy
Brief Title: Efficacy Of M-TAPA and TAP Block Following Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mursel Ekinci (Other Government)
Collaborators: Mustafa Dikici (Unknown); Ahmet Kaciroglu (Unknown)
Responsible Party: Sponsor-Investigator, Mursel Ekinci, Assoc prof, Bursa City Hospital
Organization: Bursa City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 5
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cholecystitis
Keywords: Laparoscopic Cholecystectomy; Postoperative Analgesia; Modified Perichondral Approach Thoracoabdominal Nerve Block; Transversus abdominis plane block
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Modified Perichondral Approach Thoracoabdominal Nerve block (M-TAPA block) group, and Transversus Abdominal Plane Block (TAP block) group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Modified Perichondral Approach Thoracoabdominal Nerve block group) (Active Comparator): Patients will be performed to block at the end of the surgery. Patients will be administered paracetamol 1 gr (PERFALGAN® ) IV every 8 hours in the postoperative period.. If the patient's NRS score is ≥ 4 0,5 mg/kg IV meperidine (Aldolan ampul 100 mg/2 ml) will be administered.
  Interventions: Other: Modified Perichondral Approach Thoracoabdominal Nerve block
- Group TAP (Transversus Abdominal Plane block group) (Active Comparator): Patients will be performed to block at the end of the surgery. Patients will be administered paracetamol 1 gr (PERFALGAN® ) IV every 8 hours in the postoperative period.. If the patient's NRS score is ≥ 4 0,5 mg/kg IV meperidine (Aldolan ampul 100 mg/2 ml) will be administered.
  Interventions: Other: Transversus Abdominal Plane block

INTERVENTIONS:
Other: Modified Perichondral Approach Thoracoabdominal Nerve block — M-TAPA block will be performed to Group M-TAPA at the end of the surgery, using US (Vivid Q) while the patient is in the supine position After providing aseptic conditions, the high frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed in the sagittal plane where the midclavicular line intersects with the costal cartilage corresponding to the costochondral angle. Using the In Plane technique, the probe is gently pushed to visualize the lower part of the costochondral angle at the central level, advancing the block needle in the caudal-cranio direction, 5 ml of saline will be injected into the layer between the transverse abdominal muscle and the lower plane of the costal cartilage, and the block location will be confirmed. After the block location is confirmed, a total of 20 ml + 20 ml of 0.25% bupivacaine (total 40 ml for both sides) will be injected bilaterally
  Other Names: Postoperative analgesia management
  Arms: Group M-TAPA (Modified Perichondral Approach Thoracoabdominal Nerve block group)
Other: Transversus Abdominal Plane block — TAP block will be performed to Group TAP at the end of the surgery, using US (Vivid Q) while the patient is in the supine position. After providing aseptic conditions, the high frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. USG will be placed transversely on the mid-axillary line between the iliac crest and subcostal planes. Using the In Plane technique, the block needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles and the location will be confirmed by administering 5 ml of saline. The block needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles and the location will be confirmed by administering 5 ml of saline.and than 20 ml of 0.25% bupivacaine (total 40 ml for both sides) will be injected bilaterally
  Other Names: Postoperative analgesia management
  Arms: Group TAP (Transversus Abdominal Plane block group)

SUMMARY:
Cholecystectomy is the most common abdominal surgical procedure in developed countries Laparoscopic cholecystectomy is considered the gold standard surgical technique for gallstones.

The analgesic effectiveness of TAP block has been demonstrated after laparoscopic cholecystectomy operations. m-TAPA block has been described as an alternative analgesic technique in abdominal surgeries.

The aim of this study is to compare these two analgesic methods in terms of effectiveness for postoperative analgesia management after laparoscopic cholecystectomy operations.

DETAILED DESCRIPTION:
Cholecystectomy is the most common abdominal surgical procedure in developed countries Laparoscopic cholecystectomy is considered the gold standard surgical technique for gallstones.

Several factors play a role in pain after laparoscopic cholecystectomy. This pain is complex and generally considered to be visceral. These factors are include phrenic nerve irritation caused by CO2 insufflation, abdominal distension, port incisions, the effect of gallbladder removal and individual factors.

Regional analgesia has been widely accepted by both patients and treating physicians and has become an important part of multimodal analgesia techniques. Transversus abdominis plane (TAP) block has been shown to reduce postoperative pain like hysterectomy, cholecystectomy, cesarean section and colorectal surgery.

Ultrasound (US)-guided Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) is performed by applying local anesthetic only to the underside of the perichondral surface. It provides effective analgesia in the anterior and lateral thoracoabdominal area.

M-TAPA is a good alternative for analgesia of the upper dermatome levels and lateral abdominal region and may be an opioid-sparing strategy that provides better quality recovery in patients undergoing laporoscopic surgery. M-TAPA provides analgesia at the T5-T11 level in the abdomen. Sonoanatomy is easy to visualize and the spread of local anesthetic can be easily seen with US guidance. Cephalo caudal spread of local anesthetic solution produces analgesia in several dermatomes. There are studies investigating the efficacy of M-TAPA for postoperative pain management in bariatric surgery in the literature.

Global recovery score (QoR) 15 is a sensitive, reliable and easy method to measure postoperative recovery quality. This scale, which has become a promising tool for assessing the quality of the recovery period, questions various aspects of recovery in 5 different areas: pain, physical comfort, physical independence, psychological support and emotional state. It may be an important scale to evaluate the outcome of changes in healthcare for quality assurance purposes in perioperative clinical studies. For these reasons, the "Standardized Endpoints in Perioperative Medicine" initiative and the European Society of Anesthesia have recommended the use of the QoR-15 scale in clinical studies investigating patient comfort and pain levels after surgery.

The aim of this study was to compare the efficacy of US-guided M-TAPA block and TAP for postoperative analgesia management after cholecystectomy. The primary outcome is to compare global recovery scores, the secondary outcome is to compare postoperative pain scores (NRS), to evaluate postoperative rescue analgesic (opioid) use and side effects (allergic reaction, nausea, vomiting) associated with opioid use in this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Elective laparoscopic cholecystectomy

Exclusion Criteria:

* Bleeding diathesis
* Anticoagulant treatment
* Local anesthetics and opioid allergy
* Infection at the site of block
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  The investigators will use the Turkish version of Quality of Recovery / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor])
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Patients will be evaluated at the first 24 hours period postoperatively.
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
The use of rescue analgesia | Meperidine consumption will be recorded at the first 24 hours period postoperatively.(total mg dose)
  The need for rescue analgesia will be recorded at the first 24 hours period postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Mürsel Ekinci, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Soper NJ, Stockmann PT, Dunnegan DL, Ashley SW. Laparoscopic cholecystectomy. The new 'gold standard'? Arch Surg. 1992 Aug;127(8):917-21; discussion 921-3. doi: 10.1001/archsurg.1992.01420080051008. PMID 1386505
- [Background] Donatsky AM, Bjerrum F, Gogenur I. Surgical techniques to minimize shoulder pain after laparoscopic cholecystectomy. A systematic review. Surg Endosc. 2013 Jul;27(7):2275-82. doi: 10.1007/s00464-012-2759-5. Epub 2013 Jan 24. PMID 23340814
- [Background] de Oliveira EJSG, De Lima RC, Sakata RK, Freire TT, de Almeida Lima EL, de Oliveira CMB, Moura ECR, da Cunha Leal P. Modified Thoracoabdominal Nerve Block Through the Perichondral Approach (M-TAPA) in Laparoscopic Sleeve Gastroplasty: A Case Series. Obes Surg. 2022 Jan;32(1):197-201. doi: 10.1007/s11695-021-05612-6. Epub 2021 Aug 2. No abstract available. PMID 34339018
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Myles PS, Boney O, Botti M, Cyna AM, Gan TJ, Jensen MP, Kehlet H, Kurz A, De Oliveira GS Jr, Peyton P, Sessler DI, Tramer MR, Wu CL; StEP-COMPAC Group; Myles P, Grocott M, Biccard B, Blazeby J, Boney O, Chan M, Diouf E, Fleisher L, Kalkman C, Kurz A, Moonesinghe R, Wijeysundera D. Systematic review and consensus definitions for the Standardised Endpoints in Perioperative Medicine (StEP) initiative: patient comfort. Br J Anaesth. 2018 Apr;120(4):705-711. doi: 10.1016/j.bja.2017.12.037. Epub 2018 Feb 2. PMID 29576111